CLINICAL TRIAL: NCT03582553
Title: Clinical Safety and Pharmacokinetic Evaluation of Naringenin: Single Dose Escalation Randomized Double Blind Controlled Trial
Brief Title: Safety and Pharmacokinetics of an Extract of Naringenin
Acronym: Citrus
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Collaborators: Louisiana Clinical and Translational Science Center (Other)
Responsible Party: Principal Investigator, Candida Rebello, Postdoctoral Researcher, Pennington Biomedical Research Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 2018-011
Record Dates: First submitted 2018-06-22; First posted 2018-07-11 (Actual); Results first posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Safety Issues; Pharmacokinetics
MeSH Terms: interventions — naringenin

STUDY DESIGN:
Intervention Model Description: The study consists of two cohorts of nine subjects each. In the first cohort subjects will receive the 150 mg dose and proceed to the 300 mg dose only if the 150 mg dose is deemed safe. The study is a double blind randomized controlled crossover trial, therefore, subjects could receive a placebo at the first or second visit. Similarly in the second cohort, 600 mg and 900 mg doses will be evaluated.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Except for the pharmacist who will prepare and dispense the capsules, all study staff and the investigators will be blinded to the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- 150 mg dose (Experimental): Blood will be drawn at at 0, 2, 3, 3.5, 4, 4.5, 6, 8,12, and 24 hours to measure serum naringenin concentrations in response to a single 150 mg oral dose of an extract of Citrus sinensis (sweet orange) containing naringenin and its precursor naringin.
  Interventions: Dietary Supplement: Naringenin
- 300 mg dose (Experimental): Blood will be drawn at at 0, and 4 hours to measure serum naringenin concentrations in response to a single 300 mg oral dose of an extract of Citrus sinensis (sweet orange) containing naringenin and its precursor naringin.
  Interventions: Dietary Supplement: Naringenin
- 600 mg dose (Experimental): Blood will be drawn at at 0, 2, 3, 3.5, 4, 4.5, 6, 8,12, and 24 hours to measure serum naringenin concentrations in response to a single 600 mg oral dose of an extract of Citrus sinensis (sweet orange) containing naringenin and its precursor naringin.
  Interventions: Dietary Supplement: Naringenin
- 900 mg dose (Experimental): Blood will be drawn at at 0, and 4 hours to measure serum naringenin concentrations in response to a single 900 mg oral dose of an extract of Citrus sinensis (sweet orange) containing naringenin and its precursor naringin.
  Interventions: Dietary Supplement: Naringenin
- Placebo (Placebo Comparator): Subjects in the first cohort will receive 150 mg and 300 mg ascending doses of naringenin and subjects in the second cohort will receive 600 mg and 900 mg ascending doses of naringenin. Each cohort will also have a placebo group.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Naringenin — An extract of Citrus Sinensis containing naringenin and its precursor naringin
  Arms: 150 mg dose; 300 mg dose; 600 mg dose; 900 mg dose
Other: Placebo — Cellulose
  Arms: Placebo

SUMMARY:
This study evaluates the safety of administering single ascending doses (150, 300, 600, and 900 mg) of a citrus extract of the flavonoid narigenin, and assesses the blood concentrations of naringenin following oral administration of the extract.

DETAILED DESCRIPTION:
Naringenin is a component of food with therapeutic potential to improve glucose metabolism. In order to explore the mechanisms by which naringenin may increase energy expenditure and improve glucose metabolism in humans, it is of vital importance that the safety, tolerability, and bioavailability of naringenin are evaluated, when administered to humans. This study tests the safety of four doses of a citrus extract of naringenin and measures serum concentrations of naringenin at the 150 mg and 600 mg doses over a period of 24 hours, and at the 300 and 900 mg doses at four hours after subjects have been given the respective doses of naringenin.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years)
* Body mass index between 20 and 35 kg/m2
* Must have fasting blood sugar <126 mg/dL)
* Must be willing to refrain from consuming citrus fruits and tomato in any form, for 36 hours prior to each test day.

Exclusion Criteria:

* Report citrus allergies.
* Report a history of cardiovascular disease, diabetes, or cancer
* Have evidence of hepatic disease or dysfunction
* Are currently pregnant or breastfeeding
* Are women of childbearing potential who will not use an effective method of birth control
* Chronically use of medications except over the counter medications that have been stopped 72 hours prior to the study visit
* Report clinically significant GI malabsorption syndromes
* Have clinically significant abnormal laboratory markers
* Anticipate surgery during the study period.
* Report history of substance abuse or alcoholism or significant psychiatric disorder that would interfere with the ability to complete the study.
* Have donated blood during the month prior to study entry or plan to do so during the study.
* Have participated in other studies using an investigational drug during the preceding three months.
* Are current smokers or have smoked within the previous three months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Candida Rebello, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulvihill EE, Burke AC, Huff MW. Citrus Flavonoids as Regulators of Lipoprotein Metabolism and Atherosclerosis. Annu Rev Nutr. 2016 Jul 17;36:275-99. doi: 10.1146/annurev-nutr-071715-050718. Epub 2016 May 4. PMID 27146015

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 38 subjects were screened for eligibility between May 25, 2018 and September 12, 2018.
Pre-assignment Details: Of the 38 participants screened, 10 participants did not meet the study criteria, 7 had schedule conflicts and declined to participate, and 3 were screened before the study was determined to have met the recruiting goal. 18 participants were randomized.
Groups:
- Cohort 1: NAR150, Placebo, NAR300: Cohort 1 Sequence 1: NAR150 first, then Placebo, then NAR300. 150 and 300 mg doses of naringenin where each 150 mg dose capsule (NAR150) contained 536 mg of the extract (28% naringenin determined in quantitative analysis). The 300 mg (NAR300) naringenin doses were provided in two capsules. The placebo capsules contained microcystalline cellulose and were similar in appearance.
- Cohort 1: NAR150, NAR300, Placebo,: Cohort 1 Sequence 2: NAR150 first, then NAR300 and then Placebo. 150 and 300 mg doses of naringenin where each 150 mg dose capsule (NAR150) contained 536 mg of the extract (28% naringenin determined in quantitative analysis). The 300 mg (NAR300) naringenin doses were provided in two capsules. The placebo capsules contained microcystalline cellulose and were similar in appearance.
- Cohort 1: Placebo, NAR150, NAR300: Cohort 1 Sequence 3: Placebo first, then NAR150, and then NAR300. 150 and 300 mg doses of naringenin where each 150 mg dose capsule (NAR150) contained 536 mg of the extract (28% naringenin determined in quantitative analysis). The 300 mg (NAR300) naringenin doses were provided in two capsules. The placebo capsules contained microcystalline cellulose and were similar in appearance.
- Cohort 2. NAR600, Placebo, NAR900: Cohort 2 Sequence 1: NAR600, then Placebo, and then NAR300. 600 and 900 mg doses of naringenin where each 150 mg dose capsule (NAR150) contained 536 mg of the extract (28% naringenin determined in quantitative analysis). The 600 mg (NAR600) and 900 mg (NAR900) doses of naringenin were provided in four and six 150 mg capsules respectively. The placebo capsules contained microcystalline cellulose and were similar in appearance.
- Cohort 2: NAR600, NAR900, Placebo: Cohort 2 Sequence 2: NAR600, then NAR900, and then Placebo. 600 and 900 mg doses of naringenin where each 150 mg dose capsule (NAR150) contained 536 mg of the extract (28% naringenin determined in quantitative analysis). The 600 mg (NAR600) and 900 mg (NAR900) doses of naringenin were provided in four and six 150 mg capsules respectively. The placebo capsules contained microcystalline cellulose and were similar in appearance.
- Cohort 2: Placebo, NAR600, NAR900: Cohort 2 Sequence 3: Placebo, NAR600, and then NAR300. 600 and 900 mg doses of naringenin where each 150 mg dose capsule (NAR150) contained 536 mg of the extract (28% naringenin determined in quantitative analysis). The 600 mg (NAR600) and 900 mg (NAR900) doses of naringenin were provided in four and six 150 mg capsules respectively. The placebo capsules contained microcystalline cellulose and were similar in appearance.
Period: Intervention 1/Visit 1
Arm/Group | Cohort 1: NAR150, Placebo, NAR300 | Cohort 1: NAR150, NAR300, Placebo, | Cohort 1: Placebo, NAR150, NAR300 | Cohort 2. NAR600, Placebo, NAR900 | Cohort 2: NAR600, NAR900, Placebo | Cohort 2: Placebo, NAR600, NAR900
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period ( At Least 1 Week)
Arm/Group | Cohort 1: NAR150, Placebo, NAR300 | Cohort 1: NAR150, NAR300, Placebo, | Cohort 1: Placebo, NAR150, NAR300 | Cohort 2. NAR600, Placebo, NAR900 | Cohort 2: NAR600, NAR900, Placebo | Cohort 2: Placebo, NAR600, NAR900
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention 2/Visit 2
Arm/Group | Cohort 1: NAR150, Placebo, NAR300 | Cohort 1: NAR150, NAR300, Placebo, | Cohort 1: Placebo, NAR150, NAR300 | Cohort 2. NAR600, Placebo, NAR900 | Cohort 2: NAR600, NAR900, Placebo | Cohort 2: Placebo, NAR600, NAR900
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period (At Least 1 Week)
Arm/Group | Cohort 1: NAR150, Placebo, NAR300 | Cohort 1: NAR150, NAR300, Placebo, | Cohort 1: Placebo, NAR150, NAR300 | Cohort 2. NAR600, Placebo, NAR900 | Cohort 2: NAR600, NAR900, Placebo | Cohort 2: Placebo, NAR600, NAR900
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Intervention 3/Visit 3
Arm/Group | Cohort 1: NAR150, Placebo, NAR300 | Cohort 1: NAR150, NAR300, Placebo, | Cohort 1: Placebo, NAR150, NAR300 | Cohort 2. NAR600, Placebo, NAR900 | Cohort 2: NAR600, NAR900, Placebo | Cohort 2: Placebo, NAR600, NAR900
Started | 3 | 3 | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1: NAR150, NAR300, Placebo: Cohort 1 Sequence 2: NAR150 first, then NAR300 and then Placebo. 150 and 300 mg doses of naringenin where each 150 mg dose capsule (NAR150) contained 536 mg of the extract (28% naringenin determined in quantitative analysis). The 300 mg (NAR300) naringenin doses were provided in two capsules. The placebo capsules contained microcystalline cellulose and were similar in appearance.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: NAR150, Placebo, NAR300 | Cohort 1: NAR150, NAR300, Placebo | Cohort 1: Placebo, NAR150, NAR300 | Cohort 2. NAR600, Placebo, NAR900 | Cohort 2: NAR600, NAR900, Placebo | Cohort 2: Placebo, NAR600, NAR900 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 3 | 3 | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.33 (16.36) | 48.0 (27.71) | 33 (19.05) | 37.0 (21.36) | 30.67 (17.70) | 55.33 (31.94) | 38.0 (15.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 2 | 3 | 2 | 12
  Male | 1 | 1 | 2 | 1 | 0 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 0 | 1 | 1 | 4
  White | 3 | 1 | 1 | 3 | 2 | 2 | 12
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Serum Naringenin Concentrations [Mean (Standard Deviation); unit: uM] | 0.02 (0.01) | 0.01 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0.008 (0.004)

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events Following a Single Dose of a Citrus Extract of Naringenin
Description: All adverse events will be recorded following the first administration of the study product or placebo. The study physician in consultation with the coordinator will review and determine whether a subject can be administered the next ascending dose. The cohorts will be run in series. There will be an interval of up to four weeks between the two cohorts. During this time an interim analysis will be conducted and a safety summary of adverse events for Cohort 1 will be compiled and reviewed by the investigators. Dose safety will be investigated by compiling by treatment (e.g. 150 mg dose, 300 mg dose, placebo) a list of adverse events. The frequency of these events will be counted and compared with the placebo group.
Time Frame: Adverse events were collected over approximately five weeks which included three study days and two washout periods of at least one week.
Population: Subjects who completed the study
Measure: Count of Participants; unit: Participants
Groups:
- 150 mg Dose: Blood will be drawn at at 0, 2, 3, 3.5, 4, 4.5, 6, 8,12, and 24 hours to measure serum naringenin concentrations in response to a single 150 mg oral dose of an extract of Citrus sinensis (sweet orange) containing 28% naringenin
- 300 mg Dose: Blood will be drawn at at 0, and 4 hours to measure serum naringenin concentrations in response to a single 300 mg oral dose of an extract of Citrus sinensis (sweet orange) containing 28% naringenin
- 600 mg Dose: Blood will be drawn at at 0, 2, 3, 3.5, 4, 4.5, 6, 8,12, and 24 hours to measure serum naringenin concentrations in response to a single 600 mg oral dose of an extract of Citrus sinensis (sweet orange) containing 28% naringenin
- 900 mg Dose: Blood will be drawn at at 0, and 4 hours to measure serum naringenin concentrations in response to a single 900 mg oral dose of an extract of Citrus sinensis (sweet orange) containing 28% naringenin.
Arm/Group | 150 mg Dose | 300 mg Dose | 600 mg Dose | 900 mg Dose | Placebo
Number analyzed (Participants) | 4 | 4 | 2 | 1 | 4
Participants
  Skin and Subcutaneous Tissue Disorders | 1 | 2 | 0 | 1 | 1
  Gastrointestinal | 1 | 0 | 0 | 0 | 2
  Musculoskeletal | 1 | 2 | 0 | 0 | 1
  Nervous System Disorders | 1 | 0 | 0 | 0 | 0
  Respiratory | 0 | 0 | 1 | 0 | 0
  Eye Disorders | 0 | 0 | 1 | 0 | 0

2. Secondary Outcome: Measurement of Area Under the Serum Naringenin Concentration Versus Time Curve at 150 and 600 mg Doses
Description: Blood will be drawn over a period of 24 hours following ingestion of the 150 and 600mg doses of naringenin and serum concentrations will be measured. The area under the serum concentration versus time curve will be determined.
Time Frame: 0, 2, 3, 3.5, 4, 4.5, 6, 8,12, and 24 hours
Population: Subjects who completed the study
Measure: Least Squares Mean (Standard Error); unit: (ug/mL) x hour
Arm/Group | 150 mg Dose | 600 mg Dose | Placebo
Number analyzed (Participants) | 9 | 9 | 18
(ug/mL) x hour | 18.41 (6.61) | 54.19 (6.61) | 0.08 (6.61)

3. Secondary Outcome: Measurement of Maximal Concentration of Serum Naringenin at 150 and 600 mg Doses
Description: Blood will be drawn over a period of 24 hours following ingestion of the 150 and 600mg doses of naringenin and serum concentrations will be measured. The maximal serum concentration will be determined.
Time Frame: 0, 2, 3, 3.5, 4, 4.5, 6, 8,12, and 24 hours
Measure: Mean (Standard Error); unit: ug/mL
Arm/Group | 150 mg Dose | 600 mg Dose | Placebo
Number analyzed (Participants) | 9 | 9 | 18
ug/mL | 4.29 (2.15) | 13.19 (2.15) | 0.009 (2.15)

4. Secondary Outcome: Measurement of Time to Peak Concentration of Serum Naringenin at 150 and 600 mg Doses
Description: Blood will be drawn over a period of 24 hours following ingestion of the 150 and 600mg doses of naringenin and serum naringenin concentrations will be measured. The time to peak serum naringenin concentration will be determined.
Time Frame: 24 hours
Population: Subjects who completed the study
Measure: Least Squares Mean (Standard Error); unit: hour
Arm/Group | 150 mg Dose | 600 mg Dose | Placebo
Number analyzed (Participants) | 9 | 9 | 18
hour | 3.17 (0.74) | 2.41 (0.74) | 0 (0)

5. Secondary Outcome: Measurement of Half Life of Naringenin at 150 and 600 mg Doses
Description: Blood will be drawn over a period of 24 hours following ingestion of the 150 and 600mg doses of naringenin and serum naringenin concentrations will be measured. The half life of naringenin will be determined.
Time Frame: 0, 2, 3, 3.5, 4, 4.5, 6, 8,12, and 24 hours
Population: Subjects who completed the study. The half-life uses all the pooled data to calculate an estimate of the slope (k) to determine the half-life estimate. We did not calculate the slope of each individual subject.
Measure: Number; unit: hour
Arm/Group | 150 mg Dose | 600 mg Dose | Placebo
Number analyzed (Participants) | 9 | 9 | 18
hour | 3.0 | 2.65 | 0

6. Secondary Outcome: Measurement of Apparent Oral Clearance of Naringenin at 150 and 600 mg Doses
Description: Blood will be drawn over a period of 24 hours following ingestion of the 150 and 600mg doses of naringenin and serum naringenin concentrations will be measured. The apparent oral clearance of naringenin will be determined.
Time Frame: 0, 2, 3, 3.5, 4, 4.5, 6, 8,12, and 24 hours
Population: Subjects who completed the study
Measure: Least Squares Mean (Standard Error); unit: L/hour
Arm/Group | 150 mg Dose | 600 mg Dose | Placebo
Number analyzed (Participants) | 9 | 9 | 18
L/hour | 10.21 (2.34) | 13.7 (2.34) | 0 (0)

7. Secondary Outcome: Measurement of Four-hour Concentration of Serum Naringenin at 300 and 900 mg Doses
Description: Blood will be drawn at 0 hours and 4 hours following ingestion of the 300 and 900mg doses of naringenin and serum naringenin concentrations will be measured.
Time Frame: 0 and 4 hours
Population: Subjects who participated in the study
Measure: Least Squares Mean (Standard Error); unit: uM
Arm/Group | 300 mg Dose | 900 mg Dose | Placebo
Number analyzed (Participants) | 9 | 9 | 18
uM | 10.7 (5.64) | 43.1 (5.3) | 0.3 (4.2)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over approximately five weeks which included three study days and two washout periods of at least one week.
Description: The study team employed open-ended and non-leading verbal questioning of the subject as the preferred method to inquire about adverse event occurrence. For example, appropriate questions included: "How are you feeling?", "Have you had any (other) medical problems since your last visit/contact?" The study staff established a diagnosis of the event based on signs, symptoms, and/or other clinical information. Subjects were asked about adverse events at each visit to the clinic for testing.
Arm/Group | 150 mg Dose | 300 mg Dose | 600 mg Dose | 900 mg Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/18
Other Adverse Events (participants affected / at risk) | 3/9 | 3/9 | 2/9 | 1/9 | 4/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150 mg Dose (N=9) | 300 mg Dose (N=9) | 600 mg Dose (N=9) | 900 mg Dose (N=9) | Placebo (N=18)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Itching (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cyst on Foot (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drowsiness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Visual Disturbance (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-05-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT03582553/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2018-07-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT03582553/Prot_SAP_001.pdf